CLINICAL TRIAL: NCT03311880
Title: Evaluating a Cognitive Remediation Intervention for Women During the Menopausal Transition: A Pilot Study
Brief Title: Evaluating a Cognitive Remediation Intervention for Women During the Menopausal Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Elena Ballantyne, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2950
Record Dates: First submitted 2017-10-02; First posted 2017-10-17 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Menopause
MeSH Terms: interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): There is no control group for this study. Therefore all participants receive the intervention.
  Interventions: Behavioral: Cognitive remediation

INTERVENTIONS:
Behavioral: Cognitive remediation — Participants will be taught compensatory strategies for subjective cognitive impairment in addition to learning about lifestyle modifications that are known to be beneficial on cognition.

SUMMARY:
The goal in this study is to evaluate the effectiveness of a cognitive remediation program that was designed specifically to address the concerns related to cognitive difficulties that are often reported among women in the menopausal transition. This cognitive remediation program has been created to provide our clients with an opportunity to learn more about the relation between menopause and cognitive function, to learn new strategies to enhance thinking skills (e.g., memory, attention) and to hear about lifestyle changes that are known to have a beneficial effect on mental functioning.

ELIGIBILITY:
Inclusion Criteria:

* Currently in menopausal transition
* Subjective cognitive complaints
* Presence of vasomotor menopausal symptoms (i.e., hot flashes)

Exclusion Criteria:

* Individuals with acute and severe depression
* Suicidal ideation
* Severe PTSD
* Psychosis
* Severe alcohol/substance use issues

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
change in self-reported cognitive difficulties | At the beginning of the first session and at the conclusion of the 5th session to assess change over time. That means measures will be administered 5 weeks later.
  beliefs about general memory abilities, confidence in decision-making abilities, confidence in one's ability to focus or concentrate, and high standards regarding one's cognitive performance using the Memory and Cognitive Confidence Scale (MACCS)

SECONDARY OUTCOMES:
Subjective distress | At the beginning of the first session and at the conclusion of the 5th session to assess change over time. That means measures will be administered 5 weeks later.
  Self-reported levels of stress, anxiety and depressive symptoms using the Depression Anxiety Stress Scale (DASS)
Vasomotor symptoms | At the beginning of the first session and at the conclusion of the 5th session to assess for change over time. That means measures will be administered 5 weeks later.
  hot flashes measured by the Hot Flash Interference Scale
Beliefs | At the beginning of the first session and at the conclusion of the 5th session to assess for change over time. That means measures will be administered 5 weeks later.
  perfectionistic beliefs about cognitive performance, and beliefs about the relation between aging, menopause and cognition using Likert scales for items generated by team consensus

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballantyne EC, King JP, Green SM. Preliminary Support for a Cognitive Remediation Intervention for Women During the Menopausal Transition: A Pilot Study. Front Glob Womens Health. 2021 Dec 23;2:741539. doi: 10.3389/fgwh.2021.741539. eCollection 2021. PMID 35005701